CLINICAL TRIAL: NCT05886517
Title: Transfemoral Transcatheter Aortic Valve Implementation at Hospital Without On-site Cardiac Surgery: Early Clinical Outcome in Patients With Prohibitive Surgical Risk.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AUSL Romagna Rimini (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAVI at Home
Record Dates: First submitted 2023-05-12; First posted 2023-06-02 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Evalutate all cause mortality at 30 days following TAVI
Masking Description: Nr. of all cause death patients at 30 days following TAVI/total patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAVI procedure (Experimental): Patients will be evaluated at baseline to access their eligibility for the procedure. The day of TAVI patients will be prepared for the procedures as the institution's standard practice for an invasive percutaneous endovascular procedure. During the pre hospital discharge period, patients will be monitored and will receive standard post-procedure care as judged appropriate by PI. At 30 days from the procedure a Fu visit will be made in order to access survival and adverse clinical events.
  Interventions: Device: Transfemoral transcatheter aortic valve implementation

INTERVENTIONS:
Device: Transfemoral transcatheter aortic valve implementation — ranscatheter aortic valve implantation, a percutaneous treatment for severe aortic valve stenosis, is increasingly performed worldwide. The pacemaker should be able to perform overdrive pacing which is essential to reduce cardiac output and transvalvular blood flow which are critical during balloon aortic valvuloplasty and valve deployment of the balloon- expandable valve. Minor adjustment may be needed for ideal positioning, but importantly this has to be done before valve implantation

SUMMARY:
Study design: single arm, interventional and multicenter study. The objectives are evaluate Safety and efficacy of TAVI in Department of Cardiology without on site cardiac Surgery for symptomatic severe aortic valve stenosis by expert operator team, in patients with prohibitive surgical risk. For the pilot phase, 20 patients will be enrolled. For whole study, all consecutive patients undergoing TAVI in center without CS on site will be enrolled to reach a number of about 200 patients.

ELIGIBILITY:
Inclusion Criteria:

* Senile degenerative aortic valve stenosis with echocardiography derived criteria: mean gradient > 40 mmHg or jet velocity > 4.0 m/s aortic valve area (AVA) of < 0.8 cm2 (or AVA index < 0.5 cm2/m2)
* Symptomatic due to aortic valve stenosis as demonstrated by NYHA Functional Class > = II
* Age >= 75 years old
* Patients with prohibitive risk established in the Heart Team and defined on the basis of the following clinica instrument criteria according with the Varc-2 consensus.
* High surgical risk (%, logES>20%, EuroSCORE II > 9 and STS score > 8%)
* Porcelain aorta (heavy circumferential calcification or severe atheromatous plaques that do not allow clamping.
* Hostile chest (abnormal chest wall anatomy due to severe kyphoscoliosis or other skeletal abnormalities, complications form to previous surgery, evidence of severe radiotion damege, history of multiple recurrent pleural effusions causing internal adhesions.
* Fragilty (slowness, weakness, exhaustion, wasting and malnutrition, poor endurance and inactivity, loss of independence, BMI < 20 Kg/m2 and or weight loss 5 kg/year, serum albumin < 3,5 g/dl, cognitive impairment or dementia)
* Severe liver disease/cirrosis
* Presence of a patent graft of an internal mammary artery crossing mildline and/or adherent to posterior table of sternum
* Severe pulmoary hypertension
* Severe right ventricular dysfunction
* Transfemoral access allowed
* Signature of informed consent

Exclusion Criteria:

* Tavi in case of aortic valve bioprosthesis (TAVI valve-in valve)
* controindication to femoral access
* Bicuspid aortic valve
* Instrumental characteristics, evaluated by angioTC, associated with an increased risk of major complications: severe left ventricle outflow tract or sub annular calcification, condition associated with an increased risk of rupture of the valve ring, presence of complex aortic plaques correlated with the possibility of dissection, valvular ring-coronary ostia distance < 10 mm associated with a high probability of coronary obstruction, severe aortic root dilatation or out of range aortic annulus diameters for TAVI are not complatible for safe valve implatation.

Ages: 75 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
number of all cause death patients in 30 days following TAVI/total TAVI patients | 4 weeks
  the simple size calculation is based on the primary endpoint mortality at 30 days. Considering a standard incidence of 6-7% 200 patients will be needed to demonstrate, wuth an alpha error of 5% the non inferiority of the alternative treatment compared to the standard considering a non inferiory margin of 3% such as to exclude mortaluty values higher than 10%, in relation at the upper limit of the 90% confidence interval calculated with the exact method of clopper and Pearson.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (3):
  - Ospedale Generale Regionale F Miulli, Acquaviva delle Fonti, Bari
  - AUSL Romagna Morgagni - Pierantoni Hospital, Forlì, Emilia-Romagna
  - Ospedale Santa Maria della Croci, Ravenna
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No